CLINICAL TRIAL: NCT02317406
Title: Effect of Probiotics on the Digestibility and Immunity in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biostime Institute of Nutrition and Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PEC13036
Record Dates: First submitted 2014-12-08; First posted 2014-12-16 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Gastrointestinal Tract Flora Composition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Active Comparator): Biostime probiotics sachet children's formula, 1.5g/d/sachet, administrated during the consumption of the first feeding-bottle of the day. Duration: 4 weeks
  Interventions: Drug: Biostime probiotics sachet children's formula
- Probiotics simulation (Placebo Comparator): Biostime probiotics sachet children's formula（placebo）, 1.5g/d/sachet, administrated during the consumption of the first feeding-bottle of the day. Duration: 4 weeks
  Interventions: Drug: Biostime probiotics sachet children's formula（placebo）

INTERVENTIONS:
Drug: Biostime probiotics sachet children's formula — Biostime probiotics sachet children's formula,1.5g Oral Single dose
  Arms: Probiotics
Drug: Biostime probiotics sachet children's formula（placebo） — Biostime probiotics sachet children's formula（placebo）,1.5g Oral Single dose
  Arms: Probiotics simulation

SUMMARY:
The purpose of this study is to evaluate the effect of the probiotic product on the GI tract flora composition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants;
* Single birth;
* Gestational age ≥ 37 weeks (=non-preterm infant, WHO);
* Birth weight: > 2500g
* Appropriate weight between P20-P80 in accordance with the weight percentile standards of the children ages 0 to 6 years in Shanghai urban areas at inclusion visit ;
* Aged > 4 months and < 6 months;
* Infants being exclusively formula-fed(no breast milk meal) at inclusion visit;
* No suffering of gastrointestinal diseases within 1 month (CCDC recommendations);
* Parents agreeing to use one of the recommended infant formulas (no probiotic, if with prebiotics, exclude it when there is GOS over 2g/100g or FOS inside);
* Consent form signed by at least one of the parents or by the legal tutor properly informed of the study;
* Parents able to understand the protocol requirements and to fill out the infants' diary.

Exclusion Criteria:

* Congenital illness or malformation;
* Significant pre-natal and/or post-natal disease;
* Mothers with metabolic or chronic diseases;
* Infants with allergic constitution and sensitive to the probiotics (CCDC recommendations);
* Infants with serious diseases, such as cardiovascular, cerebrovascular, liver, kidney and hematopoietic system diseases and internal secretion diseases, and those with mental disorder (CCDC recommendations);
* Infants administering other drugs during the administering of the study products, thus impossible to judge the efficacy or influencing the judgment of results (CCDC recommendations);
* Infants known to have current or previous illnesses/conditions or intervention which could interfere with the study (impacting tolerance and/or growth), such as gastrointestinal malformations, chronic diarrhoea, malabsorptive syndrome, malnutrition, congenital immunodeficiency, or major surgery, as per investigator's clinical judgment;
* Infant under oral antibiotic treatment at V1 visit and within the 4 weeks before V1
* Infants who used any medication or nutritional supplements (including probiotics, prebiotics etc, except for infant formula) in the 4 weeks preceding study start;
* Infants who have ever consumed the test product;
* Infants who have medical conditions for which a special diet other than standard (non hydrolyzed) cow's milk-based infant formula is required (such as cow's milk allergy, soy protein allergy, fish protein allergy, egg protein allergy, lactose intolerance, galactosemia);
* Currently participating or having participated in another clinical trial during the last month.
* Infants whose legal representatives have psychological or linguistic incapability to sign the informed consent form
* Reasons to presume that parents are unable to meet the study plan requirements (e.g. impossibility to contact study representatives in case of emergency, drug addiction etc.)

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Achieving the modulatory effect on the GI tract flora composition after the intervention. | From Baseline to week 4
  GI tract flora include Bifidobacterium, Lactobacillus, Clostridium perfringens, Enterococcus, Enterobacter, Bacteroides. Modulatory effect of GI tract flora composition was defined as two definitions. The first definition is that Lactobacillus and/or Bifidobacterium increases significantly, Clostridium perfringens decreases or has no change and Enterococcus, Enterobacter, Bacteroides has no obvious change. The other is that Lactobacillus and/or Bifidobacterium increases significantly, Clostridium perfringens decreases or has no change, Enterobacter and/or Enterococcus, Bacteroides increases significantly, but the amplification less than Lactobacillus/Bifidobacterium.
Change of Lactobacillus helveticuspopulations in stool | From Baseline to week 4

SECONDARY OUTCOMES:
average daily number of stools | From Baseline to week 4
Aaverage daily Infant Stool Form scores consistency | From Baseline to week 4
Average weekly Infant Stool Form scores amount | From Baseline to week 4
Average weekly Infant Stool Form scores color | From Baseline to week 4
Average daily number of crying episodes | From Baseline to week 4
Average daily duration of crying episodes | From Baseline to week 4
sIgA antibody levels in stool | From Baseline to week 4
sIgA antibody levels in saliva | From Baseline to week 4
change in infant weight | From Baseline to week 4
change in infant length | From Baseline to week 4
change in infant head circumference | From Baseline to week 4
The number of AE and SAE | From Baseline to week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China